CLINICAL TRIAL: NCT02644187
Title: Pain Relief During Photodynamic Therapy for Actinic Keratoses With a New Irradiation Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, John Paoli, MD, Assoc. Prof., Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VastraGotaland
Record Dates: First submitted 2015-12-15; First posted 2015-12-31 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Therapy, Photodynamic; Keratosis, Actinic; Pain
MeSH Terms: conditions — Keratosis, Actinic; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Left side first -Aktilite CL128 (Other): Randomized left side first with application of 5-aminolevulinic acid under occlusion during 3h. After that Aktilite CL128.
  Interventions: Device: Aktilite CL128; Drug: BF200-ALA/5-aminolevulinic acid
- Right side first -Aktilite CL128 (Other): Randomized right side first with application of 5-aminolevulinic acid under occlusion during 3h. After that Aktilite CL128.
  Interventions: Device: Aktilite CL128; Drug: BF200-ALA/5-aminolevulinic acid
- Left side first -BF-RhodoLED (Other): Randomized left side first with application of 5-aminolevulinic acid under occlusion during 3h. After that BF-RhodoLED.
  Interventions: Device: BF-RhodoLED; Drug: BF200-ALA/5-aminolevulinic acid
- Right side first -BF-RhodoLED (Other): Randomized right side first with application of 5-aminolevulinic acid under occlusion during 3h. After that BF-RhodoLED.
  Interventions: Device: BF-RhodoLED; Drug: BF200-ALA/5-aminolevulinic acid

INTERVENTIONS:
Device: BF-RhodoLED — Infrared light, with total dose of 37J/cm2.
  Arms: Left side first -BF-RhodoLED; Right side first -BF-RhodoLED
Device: Aktilite CL128 — Infrared light, with total dose of 37J/cm2.
  Arms: Left side first -Aktilite CL128; Right side first -Aktilite CL128
Drug: BF200-ALA/5-aminolevulinic acid — Prodrug applied to whole treatment area previous to illumination with either light source.

SUMMARY:
This pilot study will try to minimize the pain during exposure to a new red light source (RhodoLED®, Biofrontera Bioscience GmbH, Leverkusen, Germany) used for PDT without compromising its effect on AKs.

The study design will have an open and prospective, two-armed, split-face design. Participants with AK lesions distributed symmetrically on the scalp, forehead, cheeks, torso, back, arms and/or dorsal parts of the hands are eligible for inclusion. The purpose is to investigate if a modified irradiation protocol can lower the pain while having the same effect on AK clearance rates as compared to the standard PDT irradiation protocol.

Before any study-related procedures are performed, the participants will be thoroughly informed about the study and will be given the opportunity to ask questions. The participants will thereafter sign and date the informed consent form. This constitutes as visit 0.

On visit 1, a randomization to either the standard or the modified irradiation protocol will be performed on one side of the face/body and the other irradiation protocol will then be applied on the other side of the face/body. The participants should have AKs on two comparable sites, i.e. two cheeks, arms or dorsal parts of the hands. One side will be randomized to receive PDT with BF200-ALA and irradiation with the RhodoLED® lamp and the other side will receive BF200-ALA and the Aktilite CL-128 lamp (PhotoCure ASA, Oslo, Norway), which is the traditional lamp used at our department as mentioned above.

The treatment will be given at visit 1. During the treatment, the participants will be asked continuously, every third minute, to estimate the pain on each treatment side using the visual analogue scale, VAS, (where 0 is no pain and 10 is the worst pain imaginable). At the end of the treatment, the participants will also be asked to summarize the treatment as a whole on the VAS-scale. After visit 1, the participants will fill in a follow-up diary form with questions regarding adverse effects (AEs) during the hours and days after the treatment. The efficacy of the treatment will also be assessed at a follow-up (FU) visit, visit 2. The investigators are aiming for a non-inferior analysis, i.e. the new modified irradiation protocol should be at least as good as the standard irradiation protocol. The randomization is blinded for the investigator at the FU visit to minimize the possibility of favoring one irradiation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symmetrically distributed AKs on the scalp, forehead, cheeks, torso, back, arms and/or dorsal parts of the hands.
* Patients >18 years of age who have signed a written informed consent.

Exclusion Criteria:

* Pregnant or breast-feeding.
* Participating in other clinical study at the same time or within 30 days.
* Conditions associated with poor protocol compliance, e.g. excessive use of alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Pain assessment | Directly after PDT
  Pain is assessed on a visual analog scale from 0 to 10 (0=no pain at all, 10=worst pain imaginable). The patient assesses the pain during and after the illumination phase of PDT on both treatment sides.

SECONDARY OUTCOMES:
Effectiveness of PDT with the RhodoLED lamp | 3 months after treatment
  The effectiveness of PDT on both treatment sides will be compared at follow-up after 3 months. The clinical clearance of AK lesions will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: John Paoli, Assoc. Prof., Principal Investigator — Dep. of Dermatology, Sahlgrenska University Hospital
Locations (1):
- Dep. of Dermatology, Sahlgrenska University Hospital, Gothenburg, Sweden